CLINICAL TRIAL: NCT03395223
Title: Open Label Clinical Study to Evaluate the Safety and Efficacy of ProvayBlueTM (Methylene Blue) for the Treatment of Acquired Methemoglobinemia
Brief Title: MEthylene Blue In Patients With Acquired Methemoglobinemia
Acronym: MEBIPAM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Provepharm SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PVP-2016003; 2017-000290-37 (EudraCT Number)
Record Dates: First submitted 2017-12-18; First posted 2018-01-10 (Actual); Results first posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Acquired Methaemoglobinaemia
Keywords: Acquired Methaemoglobinemia; Methylene Blue
MeSH Terms: interventions — Methylene Blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ProvayBlue (Methylene Blue) arm (Experimental): Methylene Blue 0.5% will be administered.
  1 mg/kg will be administered intravenously over 5-30 minutes. If methemoglobin level remains above 30% or if clinical symptoms persist, give a repeat dose of up to 1 mg/kg one hour after the first dose.
  Interventions: Drug: Methylene Blue

INTERVENTIONS:
Drug: Methylene Blue — Administration of Methylene Blue to treat acquired methaemoglobinaemia
  Other Names: ProvayBlue

SUMMARY:
This is an open label, uncontrolled, Phase 4 study including 10 patients who present in hospital/urgent care setting with acquired methemoglobinemia. The population may include pediatric and adult patients (males and females of all ages are included).

The study will run in both the EU and the US. The aim of the study is to confirm safety and efficacy of ProvayBlueTM for the treatment of acquired methemoglobinemia and has been requested by the US-FDA as a Post-Marketing requirements.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric or adult patients (males and females of all ages are included) diagnosed with acquired methemoglobinemia and receiving treatment with ProvayBlue™ as per the treating physician's diagnosis and hospital standard of care.

Acquired methemoglobinemia is defined as a level of methemoglobinemia >30% or ≤30% in case of clinical symptoms (e.g. sleepiness, cyanosis, dizziness, etc.).

* Written informed consent obtained prior to any data collection (retrospective and prospective) for this study and study specific assessments.

Exclusion Criteria:

* Known severe hypersensitivity reactions to methylene blue or any other thiazine dye;
* Known deficiency in glucose-6-phosphate dehydrogenase (G6PD) due to the risk of hemolytic anemia as well as lack of therapeutic effect;
* Known deficiency in Nicotinamide Adenine Dinucleotide Phosphate Hydrogen (NADPH) reductase.
* Known use of selective serotonin reuptake inhibitors (SSRIs), serotonin and norepinephrine reuptake inhibitors (SNRIs), MonoAmine Oxidase (MAO) inhibitors or drugs metabolised via CYP isoenzymes anticipated during the treatment phase of the study.
* Women who refuse to stop breastfeeding for up to 8 days after receiving the last dose of ProvayBlueTM.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-07-06 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Megarbane, Principal Investigator — Hôpital Lariboisière
Locations (1):
- Hôpital Lariboisière, Paris, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was from July 2018- August 2020. There were 13 hospital/urgent care sites initiated in France, the United Kingdom (UK), and the United States (US).
Groups:
- ProvayBlue (Methylene Blue) Arm: Methylene Blue 0.5% will be administered.
  1 mg/kg will be administered intravenously over 5-30 minutes. If methemoglobin level remains above 30% or if clinical symptoms persist, give a repeat dose of up to 1 mg/kg one hour after the first dose.
  Methylene Blue: Administration of Methylene Blue to treat acquired methaemoglobinaemia
Period: Overall Study
Arm/Group | ProvayBlue (Methylene Blue) Arm
Started | 7
Treatment Completed | 7
Completed | 3
Not Completed | 4
Not completed — Lost to Follow-up | 3
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | ProvayBlue (Methylene Blue) Arm
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (17.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  France | 6
  United States | 1
Baseline methemoglobin [Mean (Standard Deviation); unit: percentage of methemoglobin in blood] — Percentage of methemoglobin in blood Population: One patient did not have a baseline methemoglobin result.
  percentage of methemoglobin in blood
    number analyzed (Participants) | 6
    (all) | 40.7 (21.2)

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Endpoint: Number of Participants With and Without 50% Reduction in metHb Level
Description: A 50% reduction in metHb level within 1 hour of the first dose of ProvayBlue for treatment of acquired methemoglobinemia. The timing of postdosing metHb level assays is inconsistent in clinical practice, for that reason metHb level at 1-hour postdosing was derived using linear interpolation.
Time Frame: 1 hour
Population: The efficacy analysis set includes all safety analysis set patients who have at least 1 metHb assessment before and after ProvayBlue infusion
Measure: Count of Participants; unit: Participants
Arm/Group | ProvayBlue (Methylene Blue) Arm
Number analyzed (Participants) | 6
Participants
  50% reduction in metHb level within 1 hour of the first dose: Yes | 3
  50% reduction in metHb level within 1 hour of the first dose: No | 3

2. Secondary Outcome: Number of Participants With and Without Concomitant Normalization of Respiratory Rate
Description: Normalization of the respiratory rate within 2 hours of the first dose of ProvayBlue. The normal range used for respiratory rate was 12-20 breaths per minute.
Time Frame: 2 hours
Population: All Patients who received study drug
Measure: Count of Participants; unit: Participants
Arm/Group | ProvayBlue (Methylene Blue) Arm
Number analyzed (Participants) | 7
Participants
  Respiratory rate normalized within 2 hours: Yes | 2
  Respiratory rate normalized within 2 hours: No | 2
  N/A (normal at baseline or no measurement within 2 hours of first dose) | 3

3. Secondary Outcome: Number of Participants With and Without Concomitant Normalization of Heart Rate
Description: Normalization of the heart rate within 2 hours of the first dose of ProvayBlue. The normal range used for heart rate was 50-100 beats per minute.
Time Frame: 2 hours
Population: All participants who received study drug
Measure: Count of Participants; unit: Participants
Arm/Group | ProvayBlue (Methylene Blue) Arm
Number analyzed (Participants) | 7
Participants
  Heart rate normalized within 2 hours of first dose: Yes | 2
  Heart rate normalized within 2 hours of first dose: No | 1
  N/A (normal at baseline or no measurement within 2 hours post first dose) | 4

4. Secondary Outcome: Number of Participants With and Without Concomitant Normalization of Blood Pressure
Description: Normalization of blood pressure standard values within 2 hours of the first dose of ProvayBlue. The normal range used for systolic blood pressure was was 90-140 mm HG and the normal range used for diastolic blood pressure was 60-90 mm HG.
Time Frame: 2 hours
Population: All participants who received a dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | ProvayBlue (Methylene Blue) Arm
Number analyzed (Participants) | 7
Participants
  Systolic BP: normalized within 2 hours of the first dose of ProvayBlue: Yes | 2
  Systolic BP: normalized within 2 hours of the first dose of ProvayBlue: No | 0
  Systolic BP: N/A (Normal at baseline or no measurement within 2 hours of the first dose) | 5
  Diastolic BP: normalized within 2 hours of the first dose of ProvayBlue: Yes | 0
  Diastolic BP: normalized within 2 hours of the first dose of ProvayBlue: No | 1
  Diastolic BP: N/A (Normal at baseline or no measurement within 2 hours of the first dose) | 6

5. Secondary Outcome: Second Dose
Description: Evaluation of the patients who achieve a 50% reduction in metHb level after a second dose of ProvayBlue
Time Frame: 1 hour
Population: Only 1 patient received a second dose of ProvayBlue and they did not have a metHb measurement within 1 hour of that second dose
Arm/Group | ProvayBlue (Methylene Blue) Arm
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants With Treatment-related Adverse Events
Description: Number of participants who experience a treatment emergent adverse event assessed by the investigator as being related to study drug..
Time Frame: 24 hours
Population: All participants who received at least one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | ProvayBlue (Methylene Blue) Arm
Number analyzed (Participants) | 7
Participants
  Related treatment emergent adverse event: yes | 0
  Related treatment emergent adverse event: No | 7

7. Secondary Outcome: Methylene Blue Content in Blood Samples
Description: Blood samples will be analyzed for methylene blue content
Time Frame: 24 hours
Population: Due to the nature of the disease, treatment with ProvayBlue was per the investigator's standard care and may have occurred prior to the informed consent document (PICD) being signed. However, data collection and study-specific assessments were to take place only after ICD signature. This often prevented collection of pharmacokinetic (PK) blood draws as informed consent was often given after the blood draws were to have been completed. As a result there were no patients with evaluable PK data.
Arm/Group | ProvayBlue (Methylene Blue) Arm
Number analyzed (Participants) | 0

8. Secondary Outcome: Azure B Content in Blood Samples
Description: Blood samples will be analyzed for Azure B content
Time Frame: 24 hours
Population: as for outcome 7
Arm/Group | ProvayBlue (Methylene Blue) Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AEs reported after the first dose infusion start time and within 10 days after the last dose treatment were collected.
Arm/Group | ProvayBlue (Methylene Blue) Arm
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ProvayBlue (Methylene Blue) Arm (N=7)
Thrombosis (Vascular disorders) | 1 (1) — lower limb thrombosis [right femoral vein + left fibular vein]
Methaemoglobinaemia (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study experienced a slow pace of enrollment leading to enrollment being closed prior to completing enrollment of the planned sample size of 10 subjects. Additionally, the nature of the disease and indication, necessitated that the subject's treatment with ProvayBlue was per the investigator's standard care and could have occurred prior to or after the PICD was signed. This frequently prevented the collection of pharmacokinetic (PK) blood draws and study specific evaluations on schedule.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-08-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT03395223/Prot_004.pdf
  • Statistical Analysis Plan (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT03395223/SAP_003.pdf